CLINICAL TRIAL: NCT01043289
Title: A Randomised, Double-blind, Placebo-controlled Study of Light Therapy for Antepartum Depression
Brief Title: Light Therapy for Depression During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Collaborators: Basel Women's University Hospital (Other); Columbia University (Other); University of Pittsburgh (Other); Velux Fonden (Other)
Responsible Party: Wirz-Justice, Anna / Professor, Centre for Chronobiology, Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPK-2004; 3100A0-102190/1, 320000-114110 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Major Depressive Disorder; Pregnancy
Keywords: light therapy; antepartum depression; controlled trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright light therapy (Experimental): Early morning white light @ 7,000 lux for 60 minutes daily (4.2 x 10^5 lux-min) for 5 weeks
  Interventions: Other: Light therapy
- Dim red light (Placebo Comparator): Early morning dim red light @ 70 lux for 60 minutes daily (3.0 x 10^3 lux-min) for 5 weeks
  Interventions: Other: Light therapy

INTERVENTIONS:
Other: Light therapy — During the 5-week treatment period, subjects sit in front of a light box for 60 minutes daily after awakening, at a specified distance that provides the required light intensity.
  Other Names: Phototherapy

SUMMARY:
The purpose of this study is to determine whether morning bright light therapy is an effective treatment for major depression during pregnancy compared with low-intensity placebo light therapy, when administered 60 minutes daily for 5 weeks.

DETAILED DESCRIPTION:
Affective disorder during pregnancy is a common and severe condition, associated with a higher risk for prenatal complications, preterm delivery, a higher rate of surgical birth and vaginal operative delivery. Depressed pregnant women are at risk for inadequate nutrition, poor weight gain, increased use of nicotine, drugs and alcohol, and failure to obtain adequate prenatal care, as well as poor mother-child attachment. Their infants have a higher risk for low birth weight, a higher rate of admission to neonatal intensive care, and cognitive, emotional and behavioural disturbances.Treatment of antepartum depression requires careful judgement to minimise risk to the foetus. Pharmacological treatment is an option, but all antidepressants cross the placenta, and both practitioners and patients are concerned about possible teratogenicity, pre- and perinatal adverse effects for the infant, as well as negative effects on long-term development. Thus, psychiatric medication use for depression in pregnancy may also pose an excess risk of preterm delivery and withdrawal symptoms in the newborn. Treatment of depression during pregnancy that is efficacious, reliable, safe, and with minor side effects is an urgent unmet clinical need. Light therapy may provide this somatic, non-pharmaceutical alternative. It is well established as the treatment of choice for Seasonal Affective Disorder (SAD), and there is a growing data base for response in nonseasonal major depression. Two promising pilot studies led to the present randomised, double-blind, placebo-controlled trial of 5 weeks daily morning bright light therapy (1h, 7000 lux white) compared with low-intensity placebo light therapy (1h, 70 lux red).

ELIGIBILITY:
Inclusion Criteria:

* German-speaking
* Medically healthy with normal ocular function
* Pregnancy 4 through 32 weeks gestation based on first trimester ultrasound
* DSM-IV diagnosis of major depressive disorder
* SIGH-ADS [Structured Interview Guide for the Hamilton Depression Rating Scale (HAMD) with Atypical Depression Supplement] score of >20
* Able to provide informed consent
* Preferably untreated; exception when on antidepressant for more than 3 months without any improvement, keeping medication constant during the study

Exclusion Criteria:

* DSM-IV diagnoses of bipolar 1 or 2 disorder or any psychotic episode
* Substance abuse within the last 6 months
* Primary anxiety disorder
* Recent history of suicide attempt (6 months)
* Delayed sleep phase disorder or hypersomnia with habitual sleep onset later than 1 a.m. or wakening later than 9 a.m.
* Obstetrical care or medications for medical disorders which might confound treatment results
* Fetal malformations and intrauterine fetal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change in depression ratings (HAMD, SIGH-ADS) | 5 weeks

SECONDARY OUTCOMES:
Effect of light therapy on circadian rhythms (e.g. melatonin, rest-activity cycle) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wirz-Justice, PhD, Principal Investigator — Psychiatric Hospital of the University of Basel
Locations (1):
- Psychiatric Policlinic of the University of Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Epperson CN, Terman M, Terman JS, Hanusa BH, Oren DA, Peindl KS, Wisner KL. Randomized clinical trial of bright light therapy for antepartum depression: preliminary findings. J Clin Psychiatry. 2004 Mar;65(3):421-5. doi: 10.4088/jcp.v65n0319. PMID 15096083
- [Background] Oren DA, Wisner KL, Spinelli M, Epperson CN, Peindl KS, Terman JS, Terman M. An open trial of morning light therapy for treatment of antepartum depression. Am J Psychiatry. 2002 Apr;159(4):666-9. doi: 10.1176/appi.ajp.159.4.666. PMID 11925310
- [Derived] Wirz-Justice A, Bader A, Frisch U, Stieglitz RD, Alder J, Bitzer J, Hosli I, Jazbec S, Benedetti F, Terman M, Wisner KL, Riecher-Rossler A. A randomized, double-blind, placebo-controlled study of light therapy for antepartum depression. J Clin Psychiatry. 2011 Jul;72(7):986-93. doi: 10.4088/JCP.10m06188blu. Epub 2011 Apr 5. PMID 21535997
- See also: The Center for Environmental Therapeutics is a 501(c)(3) nonprofit organization made up of a multidisciplinary team of researchers and clinicians for the development and application of effective environmental therapies — http://www.cet.org